CLINICAL TRIAL: NCT04857047
Title: A Randomized, Open-label, Multiple Doses, Crossover Clinical Study to Compare the Pharmacokinetic Characteristics and the Safety Between Administration of BR9003 and BR9003A in Healthy Adult Subjects
Brief Title: A Multi Doses Study to Compare the Pharmacokinetics of BR9003A and BR9003 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-VRNS-CT-101
Record Dates: First submitted 2021-04-09; First posted 2021-04-23 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): [Period1] administration of BR9003A 1mg twice a day for six days
  - Wash out for 9days -
  [Period2] administration of BR9003 2mg once a day for six days
  Interventions: Drug: BR9003 2mg; Drug: BR9003A 1mg
- Group B (Experimental): [Period1] administration of BR9003 2mg once a day for six days
  - Wash out for 9days -
  [Period2] administration of BR9003A 1mg twice a day for six days
  Interventions: Drug: BR9003 2mg; Drug: BR9003A 1mg

INTERVENTIONS:
Drug: BR9003 2mg — After fasting for at least 10 hours from 10:00 p.m. the previous day, one BR9003 tablet will be administered orally with 150mL of water around 8:30 a.m. after starting breakfast 30 minutes before the scheduled time of administration and finishing it.
Drug: BR9003A 1mg — After fasting for at least 10 hours from 10:00 p.m. the previous day, one BR9003A tablet will be administered orally with 150mL of water around 8:30 a.m. after starting breakfast 30 minutes before the scheduled time of administration and finishing it. Another BR9003A tablet will be administered orally with water 150mL around 20:30 after dinner between 18-19:00.

SUMMARY:
This is a randomized, multiple doses, crossover clinical study to compare the pharmacokinetic characteristics and the safety between administration of BR9003 and BR9003A in healthy adult subjects. Within each period, randomized subjects will be taken 2 dosing regimens of administrating BR9003 once a day for six days or BR9003A twice a day for six days.

DETAILED DESCRIPTION:
*Study Objective: After repeated administration of BR9003 2mg and BR9003A 1mg for healthy adult volunteers, the pharmacokinetic properties and safety are evaluated.

* Target number of subjects for enrollment (randomization):

  24 subjects in total (2 sequence groups(A or B), 12 subjects per sequence group)
* Investigational Product

  1. Control drug: BR9003A 1mg
  2. Test drug: BR9003 2mg
* Regimen

  1. Control group: Administration of BR9003A 1mg twice a day for six days
  2. Test group: Administration of BR9003 2mg once a day for six days

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 55 years at screening
2. Those who weigh at least 50 kg at the time of screening and have a calculated body mass index (BMI) within the range of 18.0 to 29.0 kg/m2
3. Determined to be eligible as subjects through physical examination and interview conducted in accordance with this protocol. In other words, those who have no congenital or chronic diseases and have no abnormal symptoms or findings based on medical examination results within the last 3 years
4. Determined to be eligible as subjects as a result of clinical laboratory tests and electrocardiography performed according to this protocol
5. Voluntarily decide to participate in the study and provide written consent to follow the study directions after listening

Exclusion Criteria:

1. Those who have clinically significant diseases or a history of the diseases associated with the cardiovascular system, respiratory system, liver, kidney, nervous system, endocrine system, blood/tumor, psychiatric diseases, or urinary system
2. Those who have hypersensitivity reactions or a history of clinically significant hypersensitivity reactions to drugs containing varenicline, or drugs containing the same class ingredients, or other drugs
3. Those with clinically significant hypotension (systolic blood pressure

   ≤ 90mmHg) or hypertension (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 95mmHg) at the time of screening
4. Those with a history of gastrointestinal diseases (e.g., Crohn's disease, ulcer, etc.) or gastrointestinal surgery (however, simple appendectomy or hernia repair are excluded) that may affect the absorption of drugs
5. Any of the following results in the screening tests

   * AST or ALT > 2 times the upper limit of the normal range
   * Total bilirubin > 2.0 mg/dL
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
6. Those who continue to drink alcohol (>21 units/week; 1 unit = 10 g = 12.5 mL of pure alcohol), or are unable to abstain from drinking during the clinical study period
7. Those who continue to smoke (>10 cigarettes/day) or cannot stop smoking during hospitalization during the clinical trial period
8. Those who have participated in another clinical trial or bioequivalence test (the last day of administration of the investigational product or bioequivalence test drug) within 6 months prior to the first administration date
9. Those who have donated whole blood within 60 days prior to the first day of administration or donated blood components (apheresis) within 30 days prior to the first day of administration or who have received a blood transfusion within 30 days
10. Those who took any prescription drugs or herbal medicines within 14 days prior to the first day of administration or any over-the-counter (OTC) drugs within 7 days prior to the first day of administration (however, if other conditions are appropriate according to the judgment of the investigator, they may participate in the clinical trial.)
11. Those who took drugs inducing and inhibiting drug-metabolizing enzymes, such as barbital, within 30 days prior to the study initiation
12. Those who have been on a diet (especially grapefruit juice or its products) that may affect the absorption, distribution, metabolism, and excretion of the drug within 7 days prior to the first day of administration
13. Pregnant woman, potentially pregnant woman, or breast-feeding woman
14. Those who do not agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy using a medically acceptable methods of contraception* throughout the entire period from the date of the first administration of the investigational product to the end of the clinical trial
15. Those who are unwilling or unable to comply with the dietary and lifestyle guidelines required for the clinical trial
16. Those who have clinically significant abnormalities in the results of other clinical laboratory tests or who have been determined by the investigator to be ineligible to participate in the clinical trial due to other reasons (e.g., non-compliance with instructions, uncooperative attitude, etc.)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
AUC0-24,ss | 0-72 hours after administration
  Area under the plasma drug concentration-time curve of BR9003 and BR9003A within 24 hours
Cmax,ss | 0-72 hours after administration
  Maximum concentration of drug in plasma of BR9003 and BR9003A within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Cho, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No